CLINICAL TRIAL: NCT01037855
Title: A Prospective Observational Study of Safety and Occurrence of Influenza-like Illness Following Administration of Adjuvanted Swine Origin A(H1N1) Pandemic Subunit Vaccine Celtura
Brief Title: Observational Study of Safety of Flu Cell Culture Derived Adjuvanted Swine Origin A (H1N1) Pandemic Subunit Vaccine
Status: Completed | Type: Observational
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: V110_07OB
Record Dates: First submitted 2009-12-20; First posted 2009-12-23 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Novel Influenza A (H1N1); A New Flu Virus of Swine Origin
Keywords: Swine Flu H1N1 vaccine; Adjuvanted flu cell culture derived

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (6):
- Group 1: 6-23 months
  Interventions: Other: Non-intervention observational study
- Group 2: 2-8 years
  Interventions: Other: Non-intervention observational study
- Group 3: 9-17 years
  Interventions: Other: Non-intervention observational study
- Group 4: 18-44 years
  Interventions: Other: Non-intervention observational study
- Group 5: 45-60 years
  Interventions: Other: Non-intervention observational study
- Group: >60 years
  Interventions: Other: Non-intervention observational study

INTERVENTIONS:
Other: Non-intervention observational study — Non-intervention observational study

SUMMARY:
This is an observational study of safety and occurrence of influenza-like illness following administration of flu cell culture derived adjuvanted swine origin A (H1N1) pandemic subunit vaccine in subjects 6 months of age and older.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 6 months
* Subjects will be vaccinated with Flu Cell Culture Derived Adjuvanted Swine Origin A (H1N1) Pandemic Subunit Vaccine, independently of this study.
* Subjects or parent/guardian willing to provide informed consent prior to vaccination administration and complete all of the study, including follow-up contact

Exclusion Criteria:

• Received any prior H1N1 vaccination

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: population of children, adolescents, adults and elderly
Sampling Method: Non-Probability Sample
Enrollment: 4028 (Actual)
Dates: Start 2009-12; Primary Completion 2010-06 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To quantify the safety of Flu Cell Culture Derived Adjuvanted Swine Origin A(H1N1) Pandemic Subunit Vaccine in actively monitored subjects | 6 months
To characterize the incidence of AEs in specific age groups following an active surveillance of vaccinated subjects | 6 months

SECONDARY OUTCOMES:
To assess the occurrence of laboratory confirmed H1N1sw and influenza-like illness following vaccination | 6 Months

CONTACTS AND LOCATIONS:
Locations (10):
- Clinica Indisa, Av. Santa Maria, Santiago Metropolitan, Chile
- Colombia (6):
  - Fundación Universitaria de Ciencias de Salud- Hospital San José Calle, Bogotá
  - Nueva EPS: Centro de Especialistas Barrios Unidos - MEDERI, Calle 66 # 40-07 - Bogotá
  - Hospital local de Yopal E.S.E, Calle 9 No. 24-37 - Yopal, Casanare
  - Clinica del Country, Carrera 16 No. 82-57 Bogotá
  - Hospital Universitario Infantil San José, Carrera 52 No. 67a-71 - Barrios Unidos - Bogotá
  - CAIMED - Centro de Atencion e Investigación Medica, Cra. 42 A No. 17-50
- Augustenburger Platz 1, State of Berlin, Germany
- Switzerland (2):
  - Policlinique Médicale Universitaire, Rue Du Bugnon 44, Ch-1011 Lausanne
  - Institute of Social and Preventive Medicine, Division of Communicable Diseases, Hirschengraben 84, Ch-8001 Zürich